CLINICAL TRIAL: NCT00237432
Title: HCV Pathogenesis and Dendritic Cell Immunobiology
Brief Title: Study of the Immune Response to Hepatitis C Virus
Status: Completed | Type: Observational
Sponsor: Rockefeller University (Other)
Responsible Party: Charles Rice, Rockefeller University
Other Study IDs: CRI-0505
Record Dates: First submitted 2005-10-10; First posted 2005-10-12 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — White blood cells
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate the mechanism of a successful immune response to hepatitis C virus (HCV) infection. Currently, it is believed that the immune system is involved in responding to HCV infection, but how it is involved is not known. It is estimated that 30% of individuals infected with HCV are able to clear the virus without treatment, while 70% progress to chronic infectious. By studying the immune responses in these two populations, we, the researchers at Rockefeller University, hope to gain insight into the mechanisms of the immune response and develop new strategies for HCV therapy.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) infects approximately 200 million people worldwide. About 30% of infected individuals do not require treatment to clear the virus, but the remainder can become chronically infected with HCV. Both resolution and protection correlate with the presence of HCV-specific T cells responses. The researchers believe that dendritic cells (DCs) play a role in determining how T-cells respond to the virus. They believe that the virus is able to modify the function of these cells causing the inactivation of T cells that would otherwise react with the virus. By characterizing the phenotype and function of DCs in both the patients who spontaneously resolve the infection and patients who become chronically infected the investigators hope to learn more about the pathogenesis of HCV.

People interested in participating in this study will have a complete history and general medical examinations before beginning the study. Testing for communicable diseases, including hepatitis B, syphilis and HIV will be done. If a disease is found you will be informed and offered counseling.

Following the screening, you will have a procedure called leukapheresis, in which white blood cells are removed, but your own red blood cells are returned. The procedure takes approximately 3 hours and is similar to blood donation. The leukapheresis is done during a same day admission to the hospital by an outside blood collection company with trained nurses and certified equipment.

Some aspects of this study are experimental which means the fluid and cells collected will be studied and analyzed to determine more precisely how your body's immune system is responding to the virus. These tests are experimental in that they are not part of the usual routine care of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed HCV infection based on serologic studies and/or plasma HCV titers
* Individuals who have recovered from toxicity of any prior therapy and who have not had IFN-α and/or ribavirin therapy in the last 6 months
* Performance status: Karnofsky 70-100%
* Life expectancy of at least 12 months
* Hematology laboratory results of:

  * WBC greater than 3,800/mm3
  * Absolute lymphocytes greater than 1,500/mm3
  * Platelets greater than 120,000/mm3
  * Hb at least 9.5 g/dl
  * INR < 1.5 IU

Exclusion Criteria:

* Patients who are currently on immunotherapy
* Individuals who are currently on antibiotics
* Individuals who have had chemotherapy within the last year for other medical conditions
* Individuals who have had corticosteroid treatment or radiotherapy within the last 4 weeks
* Individuals infected with HIV, syphilis or hepatitis B or with other serious uncontrolled medical illness
* People with currently active second malignancy other than non-melanoma skin cancer
* No history of vasculitis
* No alcohol or drug use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements
* No patients with decompensated cirrhosis
* No NYHA class III/IV status
* No severe debilitating pulmonary disease
* No psychiatric illness or social condition that, in the opinion of the investigator, would interfere with adherence to study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with confirmed HCV infection recruited from the NYC metropolitan area
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2003-04; Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles M. Rice, PHD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University Hospital, New York, New York, United States